CLINICAL TRIAL: NCT04680338
Title: Early Detection of Silent Myocardial Ischemia and Cardiac Dysfunction in Asymptomatic Individuals With Increased Coronary Artery Calcium Scores
Brief Title: Early Detection of Silent Myocardial Ischemia
Acronym: EarlySynergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pim van der Harst (Other)
Responsible Party: Sponsor-Investigator, Pim van der Harst, Clinical professor, Principal Investigator, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL64860.042.18
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Ischemic Heart Disease; Silent Myocardial Ischemia; Cardiovascular Diseases
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac magnetic resonance imaging (Active Comparator): Cardiac magnetic resonance (CMR) stress perfusion imaging with feedback of clinically actionable findings
  Interventions: Diagnostic Test: CMR stress perfusion imaging
- Control (No Intervention): No intervention, following the natural course of coronary atherosclerosis

INTERVENTIONS:
Diagnostic Test: CMR stress perfusion imaging — CMR stress perfusion imaging with feedback of clinically actionable findings to general practitioner and participant
  Arms: Cardiac magnetic resonance imaging

SUMMARY:
Early-Synergy investigates a diagnostic imaging approach in asymptomatic individuals from the general population for early detection of silent myocardial ischemia and cardiac dysfunction. The diagnostic imaging approach consists of cardiac computed tomography for coronary artery calcium scoring (CT-CAC) and cardiac magnetic resonance (CMR) stress perfusion imaging. Early-Synergy investigates the effect of early detection of silent myocardial ischemia and cardiac dysfunction by CMR in asymptomatic individuals with increased CAC. In addition, the diagnostic yield of CMR for early detection of silent myocardial ischemia and cardiac dysfunction is investigated. Asymptomatic individuals at increased risk (CAC ≥ 300) are therefore randomized 1:1 to either CMR stress perfusion imaging or a control group.

DETAILED DESCRIPTION:
Early-Synergy is a prospective multi-center study performed in the Netherlands. Potential candidates for participation in Early-Synergy have had CT-CAC scanning as part of participation in two ongoing population-based studies (ROBINSCA and ImaLife) and had CAC ≥300.

Participants are randomized in a 1:1 fashion to (1.) CMR stress perfusion imaging with feedback of clinically actionable findings or (2.) control group.

In the CMR group, feedback on CMR stress perfusion imaging is provided to the participant and general practitioner only in case of CMR findings that require further management based on current clinical guidelines. Participants in the control group will not receive stress CMR perfusion imaging but will be followed in time to evaluate the clinical presentation of the natural course of coronary atherosclerosis.

Follow-up will be performed up to 5 years in both groups by sending questionnaires and collecting medical information from health care providers and registries. Additionally, blood is drawn from participants in the CMR group during the hospital visit for CMR scanning and is stored to allow evaluation of cardiac blood markers as predictors of CMR findings.

ELIGIBILITY:
Inclusion Criteria:

* Participation in ROBINSCA or ImaLife study
* CT-CAC ≥300

Exclusion Criteria:

* History of ischemic heart disease or other cardiac disease (myocardial infarction, sudden cardiac arrest, heart failure, cardiomyopathy, congenital cardiac disease, percutaneous coronary intervention, coronary artery bypass grafting surgery, valvular surgery, other major cardiac surgery (e.g. cardiac transplantation) and/or previous invasive coronary angiography or catheter ablation)
* Contra-indication for stress CMR perfusion imaging (claustrophobia, CMR incompatible device (e.g., Implantable Cardioverter Defibrillator/pacemaker), contrast agent or vasodilator intolerance, contra-indications for adenosine or regadenoson (e.g. 2nd/3rd degree atrioventricular block, severe hypotension) and/or weight > 125 kg)
* Severe comorbidity and/or a life expectancy of less than 1 year
* Unable to provide written informed consent
* Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac events | 1 year
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
Rate of major adverse cardiac events | 2.5 years
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
Rate of major adverse cardiac events | 5 years
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
Diagnostic yield of CMR stress perfusion imaging | Baseline
  Prevalence and extent of silent myocardial ischemia and cardiac dysfunction

SECONDARY OUTCOMES:
Rate of individual components of primary outcome 1 | 1 year
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
Rate of individual components of primary outcome 1 | 2.5 years
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
Rate of individual components of primary outcome 1 | 5 years
  Cardiovascular death, non-fatal myocardial infarction or hospitalization for unstable angina, heart failure or resuscitated cardiac arrest
All-cause mortality rate | 1 year
  Death from any disease
All-cause mortality rate | 2.5 years
  Death from any disease
All-cause mortality rate | 5 years
  Death from any disease
Rate of invasive cardiovascular procedures | 1 year
  percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG) surgery, invasive coronary angiography (ICA) and other invasive cardiovascular procedures
Rate of invasive cardiovascular procedures | 2.5 years
  percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG) surgery, invasive coronary angiography (ICA) and other invasive cardiovascular procedures
Rate of invasive cardiovascular procedures | 5 years
  percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG) surgery, invasive coronary angiography (ICA) and other invasive cardiovascular procedures
Rate of hospitalization for cardiovascular disease | 1, 2.5, 5 years
  Hospitalization for cardiovascular disease (e.g. stroke, peripheral vascular disease)
Rate of hospitalization for cardiovascular disease | 1 year
  Hospitalization for cardiovascular disease (e.g. stroke, peripheral vascular disease)
Rate of hospitalization for cardiovascular disease | 2.5 years
  Hospitalization for cardiovascular disease (e.g. stroke, peripheral vascular disease)
Rate of non-invasive cardiac imaging procedures | 5 years
  Rate of non-invasive cardiac imaging procedures (e.g., myocardial stress perfusion imaing, echocardiography)
Rate of medical therapy initiation | 1 year
  Initiation of preventive or cardio-active medication (e.g., ACE-inhibiters, statins, calcium antagonists, beta-blockers etc.)
Rate of medical therapy initiation | 2.5 years
  Initiation of preventive or cardio-active medication (e.g., ACE-inhibiters, statins, calcium antagonists, beta-blockers etc.)
Rate of medical therapy initiation | 5 years
  Initiation of preventive or cardio-active medication (e.g., ACE-inhibiters, statins, calcium antagonists, beta-blockers etc.)
Quality of Life as reflected by EQ-5D-5S score | 1 year
  Quality of life as assessed by EQ-5D-5S questionnaire
Quality of Life as reflected by EQ-5D-5S score | 2.5 years
  Quality of life as assessed by EQ-5D-5S questionnaire
Quality of Life as reflected by EQ-5D-5S score | 5 years
  Quality of life as assessed by EQ-5D-5S questionnaire
Quality of Life as reflected by HeartQoL score | 1 year
  Quality of life as assessed by HeartQoL questionnaire
Quality of Life as reflected by HeartQoL score | 2.5 years
  Quality of life as assessed by HeartQoL questionnaire
Quality of Life as reflected by HeartQoL score | 5 years
  Quality of life as assessed by HeartQoL questionnaire

OTHER OUTCOMES:
Cost-effectiveness | 1 year
  Cost-effectiveness of CMR stress perfusion imaging compared to control group
Cost-effectiveness | 2.5 years
  Cost-effectiveness of CMR stress perfusion imaging compared to control group
Cost-effectiveness | 5 years
  Cost-effectiveness of CMR stress perfusion imaging compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: Pim van der Harst, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data management plan in progress
Supporting Information: Study Protocol, SAP
Time Frame: In accordance with legal period for study data storage
Access Criteria: In correspondence with the principal investigator

REFERENCES:
- [Background] Xia C, Rook M, Pelgrim GJ, Sidorenkov G, Wisselink HJ, van Bolhuis JN, van Ooijen PMA, Guo J, Oudkerk M, Groen H, van den Berge M, van der Harst P, Dijkstra H, Vonder M, Heuvelmans MA, Dorrius MD, De Deyn PP, de Bock GH, Dotinga A, Vliegenthart R. Early imaging biomarkers of lung cancer, COPD and coronary artery disease in the general population: rationale and design of the ImaLife (Imaging in Lifelines) Study. Eur J Epidemiol. 2020 Jan;35(1):75-86. doi: 10.1007/s10654-019-00519-0. Epub 2019 Apr 23. PMID 31016436
- [Background] Vonder M, van der Aalst CM, Vliegenthart R, van Ooijen PMA, Kuijpers D, Gratama JW, de Koning HJ, Oudkerk M. Coronary Artery Calcium Imaging in the ROBINSCA Trial: Rationale, Design, and Technical Background. Acad Radiol. 2018 Jan;25(1):118-128. doi: 10.1016/j.acra.2017.07.010. Epub 2017 Aug 23. PMID 28843465